CLINICAL TRIAL: NCT05493332
Title: A Prospective, Single-armed, Multicentric, Explorative Phase II Clinical Research of Conversional Therapy With Combination of Hepatic Arterial Infusion Chemotherapy and Donafenib and Toripalimab for Unresectable Hepatocellular Carcinoma
Brief Title: HAIC Combined With Donafenib Tosilate and Toripalimab for Unresectable HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-128
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; toripalimab; donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC-Donafenib-Toripalimab Group (Experimental): HAIC(FOLFOX)+Toripalimab+Donafenib
  Interventions: Procedure: HAIC(FOLFOX); Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Toripalimab; Drug: Donafenib

INTERVENTIONS:
Procedure: HAIC(FOLFOX) — After successful percutaneous hepatic artery cannulation, superior mesenteric arteriogram and hepatic arteriogram were performed, and after confirming that the subjects were eligible for enrollment according to the results, the hepatic artery was cannulated to the predetermined position. The catheter was connected to a syringe pump in the ward for continuous pumping of chemotherapy drugs.
  Other Names: Hepatic Artery Infusion Chemotherapy; FOLFOX
Drug: Oxaliplatin — 85mg/m2 IVdrip from hour 0 to 2 on D1，Q3W
Drug: Leucovorin — 400mg/m2 IVdrip , from hour 0 to 2 on D1 to D2，Q3W
Drug: Fluorouracil — 400mg/m2 , bolus at hour 3 ; and 600mg/m2 IVdrip over 46 hours on D1 to D2，Q3W
Drug: Toripalimab — 240mg IVdrip，D3, Q3W
Drug: Donafenib — 0.1g. P.O, BID, continuously

SUMMARY:
This is a prospective, single-armed, multicentric, explorative phase II clinical research of conversional therapy with combination of hepatic arterial infusion chemotherapy(HAIC), Donafenib Tosilate and Toripalimab for unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Compared with systemic intravenous chemotherapy, hepatic arterial infusion chemotherapy(HAIC) has the advantages of increasing local drug concentration and reducing systemic toxic and side effects. Currently, it is gradually used in the treatment of hepatocellular carcinoma (HCC) with good safety and high objective response rate. Immunotherapy combined with targeted and chemotherapy was well tolerated. At present, anti-programmed cell death protein-1(PD-1) antibody combined with chemotherapy and targeted therapy for advanced biliary tract tumors has initially shown good safety and encouraging efficacy, which is worthy of further exploration. Therefore, this study aims to evaluate the efficacy and safety of HAIC (FOLFOX) combined with Toripalimab and Donafenib Tosilate in unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent form, abled to comply with visits and related procedures specified in the program;
* Age 18-75 years old (including the boundary value), male or female;
* Zubrod-ECOG-WHO scored 0 to 1;
* Expected survival time ≥ 12 weeks;
* Serum AFP detection and imaging examination meet the clinical diagnostic criteria for hepatocellular carcinoma in the "National Health Commission of the People's Republic of China. Guidelines for diagnosis and treatment of primary liver cancer in China (2019 edition)";
* Liver function grading: Child-Pugh grade A or better B grade (≤7 points);
* According to the modified solid tumor efficacy evaluation criteria (mRECIST), at least one imaging measurable lesion;
* Newly diagnosed hepatocellular carcinoma patients who have not undergone any local or systematic treatment for hepatocellular carcinoma in the past;
* Patients with hepatocellular carcinoma who have been evaluated by researchers and do not have the conditions for radical resection surgery, but are expected to achieve radical resection through translational therapy, include but are not limited to one of the following situations:

  1. The tumor is massive, close to or involves the main intrahepatic ducts, and the surgical margin is expected to be 1 cm or closer to the edge of the tumor, making it difficult to achieve R0 resection;
  2. The tumor is large, but limited to the target resection of the liver segment;
  3. Tumors with large vascular carcinoma suppositories, such as portal vein primary branch carcinoma suppositories (not entering the main trunk), hepatic vein cancer suppositories (not entering the inferior vena cava), but portal vein cancer embolus can only be limited to one side and cannot affect the contralateral side;
  4. Tumor nodules ≥ 4, and mainly concentrated on the side of the liver;
  5. other conditions in which the researcher believes that radical resection may be achieved through translational therapy;
* Full organ and bone marrow function, and the laboratory test values within 7 days before enrollment meet the following requirements (no blood components, cell growth factors, albumin, and other drugs for corrective treatment are allowed within the first 14 days of obtaining laboratory tests), as follows:

  1. Blood count: absolute neutrophil count (ANC) ≥ 1.5×10^9/L; Platelet count (PLT) ≥75×10^9/L; Hemoglobin content (hemoglobin, HGB) ≥80g/L;
  2. Liver function: serum total bilirubin (TBIL) ≤ 1.5× upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransase (AST) ≤5×ULN; Serum albumin ≥ 28 g/L; alkaline phosphatase (ALP) ≤5×ULN;
  3. Renal function: serum creatinine (creatinine, Cr) ≤ 1.5× ULN or clearance of creatinine (CCr) ≥ 45mL/min (Cockcroft-Gault formula); Urinalysis results show urine protein <2+;
  4. Coagulation function: the international normalized ratio (INR) is ≤2, and the activated partial thromboplastin time (APTT) ≤ 1.5 times ULS;
  5. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) in the normal range. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
  6. Myocardial enzyme profile is within the normal range (if the researcher comprehensively judges that it is not clinically significant as a simple laboratory abnormality, it is also allowed to enroll);
* Female subjects of childbearing age should undergo a negative urine or serum pregnancy test within 7 days prior to receiving the first study drug administration (day 1 of the first cycle). If the results of the urine pregnancy test cannot be confirmed as negative, a blood pregnancy test is required. Women of non-reproductive age are defined as at least 1 year after menopause, or have undergone surgical sterilization or hysterectomy;
* If there is a risk of conception, all subjects (whether male or female) should use contraception with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last study drug administration of treatment.

Exclusion Criteria:

* Histology contains fibroblast hepatocellular carcinoma, sarcoma-like hepatocellular carcinoma, cholangiocarcinoma and other components;
* Patients with hepatocellular carcinoma who have previously undergone radical resection and recurrent hepatic cancer;
* Have received liver transplantation in the past;
* Have previously received systemic therapy for hepatocellular carcinoma, including targeted drug therapy such as sorafenib, renvatinib, and rigofenib, or immunomodulatory agent therapy such as anti-PD-1, anti-PD-L1/L2, and anti-CTLA-4, excluding antiviral therapy; If the patient has previously used Chinese medicine with anti-tumor indications, he or she must be > 2 weeks or 5 drug half-lives (whichever is longer) after the completion of treatment and before the use of this study;
* Before starting treatment, there has not been sufficient recovery from toxicity and / or complications caused by any intervention (i.e., ≤ grade 1 or reach baseline, excluding fatigue or hair loss);
* Patients with any extrahepatic organ or lymph node metastases, including but not limited to: lung metastases, bone metastases, brain metastases or local lymph node metastases;
* There are tumors in the left and right liver lobes, such as diffuse multiple tumors of the whole liver, tumor infiltration of contralateral phylloscopic vein branches, and concomitant inferior vena cava cancer suppositories, etc. There is no potential possibility of transformable resection;
* There is difficult to control hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion or pericardial effusion;
* Active bleeding or coagulation abnormalities, bleeding tendencies, or receiving thrombolytic, anticoagulant, or antiplatelet therapy;
* Major surgical procedures (craniotomy, thoracic or abdominal opening) or unhealed wounds, ulcers, or fractures that have not healed within 4 weeks prior to the first dose. Tissue aspiration biopsy or other minor surgical procedures within 7 days prior to the first administration, with the exception of a venipuncture catheter for the purpose of intravenous infusion;
* History of gastrointestinal bleeding within the previous 4 weeks or a clear tendency to bleed from the gastrointestinal tract (e.g., known focal active ulcer lesions, fecal occult blood++, gastroscopy if persistent fecal occult blood +), or other conditions determined by the researcher that may cause gastrointestinal bleeding (e.g., severe floor/esophageal varices);
* History of any arteriovenous thrombosis, embolism or ischemia in the previous 6 months, such as myocardial infarction, unstable angina, deep vein thrombosis, pulmonary embolism, cerebrovascular accident or transient ischemic attack;
* History of gastrointestinal perforation, abdominal fistula or abdominal abscess within the previous 6 months;
* Patients with past and current objective evidence of a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, and severe impairment of lung function;
* Previously or currently suffering from congenital or acquired immunodeficiency diseases;
* Active autoimmune diseases requiring systemic therapy or a history of the disease within the previous 2 years (vitiligo, psoriasis, alopecia, or Grave's disease that do not require systemic treatment within the last 2 years, hypothyroidism requiring thyroid hormone replacement therapy only, and patients with type I diabetes who require only insulin replacement therapy can be selected). Known history of primary immunodeficiency. Only patients with positive autoimmune antibodies need to be confirmed as to whether an autoimmune disease is present according to the investigator's judgment;
* Immunosuppressive drugs have been used within the previous 4 weeks, excluding nasal spray, inhalation or other routes of local glucocorticoids or physiological doses of systemic glucocorticoids (i.e., not more than 10 mg/day prednisone or equivalent doses of other glucocorticoids), allowing the temporary use of glucocorticoids for the treatment of symptoms of dyspnea in the treatment of asthma, chronic obstructive pulmonary disease and other diseases;
* Attenuated live vaccines were received within the previous 4 weeks or planned for the duration of the study；
* Other malignancies are diagnosed within 5 years prior to the first dose, excluding radically cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ. If other malignant tumors are diagnosed more than 5 years before administration, pathological or cytological diagnosis of intrahepatic lesions is required to determine whether the original malignancy is a recurrence of liver metastasis;
* Pregnant or lactating women, as well as women with fertility or male patients who are unwilling or unable to use effective contraception;
* Untreated active hepatitis B (defined as HBsAg-positive simultaneous detection of HBV-DNA copies greater than the upper limit of normal in the laboratory at the site) Note: Hepatitis B subjects who meet the following criteria can also be enrolled: 1) HBsAg (+) and/or HBcAb (+) before first administration, especially HBV replication is active (HBV-DNA≥1000copies/ml or 2000IU/ml), subjects should receive anti-HBV therapy throughout the duration of the study treatment; 2) For subjects with HBcAg (+) and HBsAg(-), HBsAg(-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring for viral reactivation is required;
* Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower detection limit);
* There are any serious or uncontrollable systemic disorders, such as: 1) Have grade II myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval male ≥ 450 ms, female ≥ 470 ms) 2) According to NYHA standard III. to IV. cardiac insufficiency or cardiac color ultrasound examination: LVEF (left ventricular ejection fraction) < 50% 3) Unsatisfactory blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure >90 mmHg); 4) Poor control of diabetes mellitus (fasting blood glucose (FBG) >10mmol/L); 5) Urine routine indicates urine protein ≥++, and confirms that the quantitative > of urine protein in 24 hours is 1.0 g; 6) Patients with mental disorders who cannot cooperate with treatment;
* Medical history or disease evidence that may interfere with test results, prevent participants from participating in the study throughout the study, abnormal treatment or laboratory test values, or other circumstances that the investigator deems unsuitable for enrolment The investigator considers other potential risks to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Conversion therapy success rate | through study completion, an average of 2 year
  Defined as the proportion of patients who met the resection criteria after conversion therapy and successfully underwent radical resection surgery to the total number of patients enrolled.

SECONDARY OUTCOMES:
Conversion therapy success rate based on imageological examination | through study completion, an average of 2 year
  Defined as the proportion of patients who met the resection criteria based on imageological proof after conversion therapy to the total number of patients enrolled.
Objective response rate (ORR) | through study completion, an average of 2 year
  Defined as proportion of patients who have a best response of treatment.
Disease control rate(DCR） | through study completion, an average of 2 year
  Defined as the proportion of cases with remission and stable lesions after treatment was assessable.
Progression-free survival（PFS） | through study completion, an average of 2 year
  Defined as the time from the date of enrollment until the date of objective disease progression or death (by any cause in the absence of progression).
Overall survival(OS) | through study completion, an average of 2 year
  Defined as time from the start of treatment until death due to any reason.
Recurrence-free survival(RFS) | through study completion, an average of 2 year
  Defined as the time from date of randomization until the date of recurrence.
Time to response（TTR） | through study completion, an average of 2 year
  Defined as the time from date of randomization until the date of patients who met a reasonable response to treatment.
Safety and tolerability（Adverse Events） | through study completion, an average of 2 year
  Safety as measured by number and grade of adverse events
Patient reported outcome（PRO） | through study completion, an average of 2 year
  Any potential types of measurement self-reported by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyu Xiao, Principal Investigator — Department of Hepatobiliary Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JW, Chen M, Colombo M, Roberts LR, Schwartz M, Chen PJ, Kudo M, Johnson P, Wagner S, Orsini LS, Sherman M. Global patterns of hepatocellular carcinoma management from diagnosis to death: the BRIDGE Study. Liver Int. 2015 Sep;35(9):2155-66. doi: 10.1111/liv.12818. Epub 2015 Mar 25. PMID 25752327
- [Background] He MK, Le Y, Li QJ, Yu ZS, Li SH, Wei W, Guo RP, Shi M. Hepatic artery infusion chemotherapy using mFOLFOX versus transarterial chemoembolization for massive unresectable hepatocellular carcinoma: a prospective non-randomized study. Chin J Cancer. 2017 Oct 23;36(1):83. doi: 10.1186/s40880-017-0251-2. PMID 29061175
- [Background] Gourd K, Lai C, Reeves C. ESMO Virtual Congress 2020. Lancet Oncol. 2020 Nov;21(11):1403-1404. doi: 10.1016/S1470-2045(20)30585-4. Epub 2020 Sep 24. No abstract available. PMID 32979983
- [Background] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690
- [Background] Bersanelli M, Buti S. From targeting the tumor to targeting the immune system: Transversal challenges in oncology with the inhibition of the PD-1/PD-L1 axis. World J Clin Oncol. 2017 Feb 10;8(1):37-53. doi: 10.5306/wjco.v8.i1.37. PMID 28246584
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338